CLINICAL TRIAL: NCT06252597
Title: Education and Training for Wheelchair Users and Caregivers for Pressure Relief Performance and Barrier Management
Brief Title: Pressure Relief Education and Training for Wheelchair Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00107536
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-11

CONDITIONS: Pressure Area
Keywords: wheelchair users; complex power wheelchairs; progressive disorders
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Clients with neuro-progressive disorders (ALS, multiple sclerosis, Parkinson's, muscular dystrophies, and spinal muscular atrophy) who also use complex power wheelchairs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- education and training (Experimental): After implementation of the pre-interview and determination/performance of necessity, education and training at a regularly scheduled occupational therapy clinic visit will be performed with handouts, verbal education, hands-on training, and video training.
  Interventions: Behavioral: education and training

INTERVENTIONS:
Behavioral: education and training — education and training at a regularly scheduled occupational therapy clinic visit will be performed with handouts, verbal education, hands-on training, and video training

SUMMARY:
There can be barriers for clients with progressive disorders who are power wheelchair users and their caregivers that prohibit them from performing pressure relief. Clients may struggle with consistent performance of pressure relief and may not recall the importance, have methods to perform, or be able to perform due to weakness or other disease changes.

DETAILED DESCRIPTION:
Study the population of power wheelchair users with progressive disorders at the Neurology Specialty Care - Edgehill, Carolina Neuromuscular Amyotrophic Lateral Sclerosis (ALS)/ Muscular Dystrophy Association (MDA) Center to identify barriers, provide potential solutions, and provide education and training to both increase knowledge and understanding of pressure relief options and processes as well as to overcome these perceived barriers amongst the clinic population. Current adults of the Neurology Specialty Care practice who are complex power wheelchair users will be eligible for this project as an extension of usual care.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older
* Diagnosis of a progressive disorder (amyotrophic lateral sclerosis (ALS), multiple sclerosis (MS), muscular dystrophy (MD), spinal muscular atrophy (SMA), Parkinson disease (PD)
* Current clinic client at the Neurology Specialty Care Edgehill clinic
* Currently using a complex (group 3) power wheelchair with power positioning of at least tilt/recline
* Currently sitting in the chair at least 2 consecutive hours/day

Exclusion Criteria:

* Dementia as noted by Medical Doctor / speech-language pathologists (SLP) in medical records
* Inability/unwillingness to control wheelchair power features (client)
* Unwillingness to be monitored, educated, trained by study staff
* Uses other mobility devices indoors (scooter, basic power wheelchair) more than complex power wheelchair
* Further exclusions may be added in future protocol versions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Likert Pain Scale Scores | Baseline
  0: Relaxed and comfortable. 1 to 3: Mild discomfort. 4 to 6: Moderate pain. 7 to 10: Severe discomfort/pain - higher scores equaling more discomfort/pain
Likert Pain Scale Scores | Week 4
  0: Relaxed and comfortable. 1 to 3: Mild discomfort. 4 to 6: Moderate pain. 7 to 10: Severe discomfort/pain - higher scores equaling more discomfort/pain
Standard Staging for any Pressure Injuries | Baseline
  Stage 1 pressure injuries are not open wounds Stage 2 pressure injuries are open wounds Stage 3 pressure injuries extend through the skin into deeper tissue and fat but do not reach muscle, tendon, or bone Stage 4 pressure injuries extend to muscle, tendon, or bone Higher scores equaling worse condition
Standard Staging for any Pressure Injuries | Week 4
  Stage 1 pressure injuries are not open wounds Stage 2 pressure injuries are open wounds Stage 3 pressure injuries extend through the skin into deeper tissue and fat but do not reach muscle, tendon, or bone Stage 4 pressure injuries extend to muscle, tendon, or bone Higher scores equaling worse condition

CONTACTS AND LOCATIONS:
Overall Officials: Amber L Ward, MS, OTR/L, Principal Investigator — Carolinas Neuromuscular ALS/MDA Center
Locations (1):
- Carolinas Neuromuscular ALS/MDA Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT06252597/ICF_000.pdf